CLINICAL TRIAL: NCT06317961
Title: Pilot Study on the Use of iENTER, iCONSENT and iPARTICIPATE E-tools
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Vall d'Hebron Institute of Oncology (Other); The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: INT200-22
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Precision oncology is the future of fighting cancer. Cancer Core Europe (CCE) developed a precision medicine trial, i.e. the Basket of Basket (BoB) study, to provide personalised treatment to a large number of patients by incorporating a molecular profiling platform. The EU-funded CCE_DART project, developed within the CCE Consortium, is aimed at improving efficiency and transform platform trials into data-rich translational research programmes. Within the CCE_DART project working area D "Patient involvement through information and partnership" three interconnected web e-tools were developed aimed at promoting patient information, recruitment, and involvement as well as facilitating adherence to the CCE BoB trial: 1) iENTER: informative web site addressed to potential BoB trial participants, their caregivers, patients' advocates, and the public; 2) iCONSENT: web app for remote management of the informed consent process in the CCE BoB trial.3) iPARTICIPATE: web app allowing remote access to BoB trial patients trial visits calendar, medications list and posology, to upload documents and download reports, messaging between patients and clinical staff. The main objective of this study is to carry out field testing and assess usability of the e-tools iENTER, iCONSENT and iPARTICIPATE. The study is also addressed at collecting patients' suggestions for improvements of the e-tools.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients, or their informal caregivers, candidates to precision oncology trials. Patients or caregivers able to surf the internet and to fill in a simple online form.

Exclusion Criteria:

* People with clinically evident cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in the CCE BoB trial
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
SUS questionnaire | 31-1-2025
  The SUS questionnaire consists of 10 Likert type items with five response options (from Strongly agree to Strongly disagree).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This website provides information that may be helpful in the process of decision making about clinical trial participation. It is targeted to patients and/or their caregivers, but it can also be used by the general public. — https://dart.datariverweb.com/iEnter/?lang=it
- See also: Building Data Rich Clinical Trials CCE_DART is an innovative EU-funded project dedicated to deliver novel methods for the design and implementation of newer, more efficient and effective clinical trials in oncology — https://cce-dart.com/